CLINICAL TRIAL: NCT05198882
Title: Clinical Evaluation of Interstitial Laser Thermal Therapy Under Continuous MRI Monitoring as a Minimally Invasive Treatment of Patients With Medically Unbalanced Partial Epilepsy
Acronym: EPILITT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP200097
Record Dates: First submitted 2021-12-06; First posted 2022-01-20 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-07

CONDITIONS: Drug-resistant Focal Epilepsy; Epilepsy; Epilepsies, Focal; Focal Epilepsy; Drug Resistant
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LITT technology (Experimental): Laser-induced thermocoagulation of intracerebral lesions responsible for drug-resistant epilepsy.
  Interventions: Procedure: Laser technology for intracerebral thermocoagulation

INTERVENTIONS:
Procedure: Laser technology for intracerebral thermocoagulation — One intervention : LITT (Laser Interstitial Thermal Treatment), technology that uses laser energy to thermally destroy (photo-thermal treatment) a brain injury under continuous MRI control (Validated by FDA - CE marking). The operator console + surgical laser generator + software that manages the power delivered by the laser is connected to an MRI - Provided by MEDTRONIC - FDA approved and CE certified.

SUMMARY:
Laser Induced Interstitial Thermal Therapy (LITT) is a "minimally invasive" procedure that uses the heat generated by a laser light (65°) to destroy brain lesions by coagulation leading to lesion necrosis under real-time MRI monitoring. The laser optical fiber is implanted into the lesion using stereotaxy. This technique, which can be performed under local anesthesia and on an outpatient basis, proved its efficacy and safety in the treatment of brain metastases for the first time in the world in 2006 (A. Carpentier et al, 2008, 2011). Since then, more than 5,000 patients have been treated in the USA, including for epileptogenic lesions (FDA device and CE cleared). Our goal is to evaluate LITT on lesions with drug-resistant epilepsy for which surgical resection is impossible. No therapeutic trial evaluating LITT in this indication has been performed to date. It is therefore necessary to study its feasibility and tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and < 80 years
2. Patient with a medically unbalanced partial epilepsy
3. Patient with a lesional image(s) in morphological MRI responsible for epilepsy based on clinical and electrophysiological assessment, +/- PET +/- SPECT +/- MEG +/- sEEG
4. Patients for whom scheduled neurosurgical treatment with craniotomy appears difficult: Deep lesions, eloquent region lesions, patient reluctance to perform surgery.
5. Endorsement of the Multidisciplinary Meeting of Neuro-epileptology
6. Patient affiliated with a social security scheme
7. Patient who has signed prior, free and informed consent

Exclusion Criteria:

1. Pharmacosensitive epilepsy
2. Patient with poor adherence to medication, or with psychological disorders
3. Patients under legal protection
4. Patient with a contraindication to MRI (metal shards, known allergy to gadolinium, etc.)
5. Anticoagulant and antiplatelet therapy underway, cannot be stopped.
6. Severe and unbalanced psychiatric disorders
7. Pregnant women. Women of childbearing age should use oral contraception throughout the study.
8. Allergy to local anaesthetics / general anaesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of post-surgical complication of grade greater or equal to 2 according to Mathon and al classification | Day 30 post-operative
  To assess the safety and feasibility of laser-induced thermocoagulation of intracerebral lesions responsible for drug-resistant epilepsy.

SECONDARY OUTCOMES:
Seizure freedom evaluated with Engel classification | Post surgery : Month 1, Month 3, Month 6, Month 12
  Evaluate the clinical epileptic efficacy of treatment based by the ILAE and Engel classifications.
Seizure freedom evaluated with ILAE (International League Against Epilepsy) classification | Post surgery : Month 1, Month 3, Month 6, Month 12
  Evaluate the clinical epileptic efficacy of treatment based by the ILAE and Engel classifications.
Number of seizure per patient | Post surgery : Month 1, Month 3, Month 6, Month 12
  Evaluate the frequency of seizure
Number of patient with at least one seizure with complex partial seizure | Post surgery : Month 1, Month 3, Month 6, Month 12
  Evaluate the intensity of seizure after treatment.
Number of patient at least one modification of anti-epileptic treatment | Post surgery : Month 1, Month 3, Month 6, Month 12
  Evaluation of clinical efficacy of treatment
Mean change of quantification of the number of interictal peaks over 30 minutes evaluated at surface EEG compared to the pre surgery surface EEG | Post surgery : Month 3, Month 6, Month 12
  Electrophysiological epileptic efficacy
Mean change neuropsychological scores | Post surgery : Month 12
  Evaluate the effect on cognition by a postoperative neuropsychological evaluation, compared with the pre-treatment neuropsychological evaluation.The neuro-psychological test will be selected according to the location of the lesion/focus
Mean change in Quality of Life in Epilepsy (QOLIE-31) scores | Post surgery : Month 6, Month 12
  Evaluate the effect on quality of life by comparing the preoperative assessment with the postoperative assessments.
Incidence of adverse events | Day of surgery, Day 2, Day 7, Day 30 post-operative
  Evaluate the clinical tolerance of the procedure.
Mean consumption of anti-epileptic drugs and epilepsy-related care | Post surgery : Month 12
  To assess the medico-economic impact of the treatment
Mean of major and minor axis measurements evaluated by measuring post-treatment morphological MRI images corresponding to induced necrosis in T1 gadolinium SPGR MRI | Month 1, Month 3, Month 12
  Evaluate the radiological epileptic efficacy of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France